CLINICAL TRIAL: NCT06426914
Title: Effect of Clinical Pilates (CP) Exercises on Kinesiophobia and Post-operative Cardiopulmonary Parameters in CABG Patients.
Brief Title: Clinical Pilates (CP) Exercises and Kinesiophobia in CABG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rec/01818 Sarosh Gohar
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Post-cardiac Surgery
Keywords: CABG; Clinical Pilates; Kinesiophobia; Post-operative cardiopulmonary parameters
MeSH Terms: conditions — Kinesiophobia | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Pilates Clinical (Introductory program)
  Interventions: Other: Clinical Pilates
- Control (Active Comparator): Cardiac Rehabilitation
  Interventions: Other: Cardiac Rehabilitation

INTERVENTIONS:
Other: Clinical Pilates — Warmup: 5-10 minutes Pilates Clinical (Introductory program) The Hundred modified The Roll-up modified The roll-over modified Spine twist modified Single-leg circle modified Rolling like a ball Shoulder Bridge modified
  For every Step emphasizing:
  FOCUS: On muscle involved REPETITIONS: 3-5 VISUALIZATION: Imagination process (Different for each step) Cool down: 5 minutes Total Time: 30 minutes
  Arms: Interventional
Other: Cardiac Rehabilitation — Chest Physical therapy (Chest percussions and active huffs as per need) Breathing strategies (Diaphragmatic and purse lip 1-3 sets * 5 Reps/Day)
  Functional mobility (walk /cycling as per patient tolerance)
  Patient education and Wound care Sternal Precaution guidance
  Arms: Control

SUMMARY:
To determine Effect of Clinical Pilates (CP) exercises on kinesiophobia and post-operative cardiopulmonary parameters in CABG patients. Kinesiophobia may lead to patients' psychological fear of rehabilitation exercise, thereby refusing rehabilitation exercise, affecting the rehabilitation process of patients, resulting in disuse syndrome, depression, disability and other adverse consequences. Thus, this study is to be conducted to find out the effects Pilates exercises with cardiac rehabilitation for management of Kinesiophobia in post CABG patients.

DETAILED DESCRIPTION:
Clinical Pilates are also evident to be safe and effective in post-surgical patients with different surgical interventions.

A study was conducted in 2021 to evaluate the effects of the Pilates method on pulmonary function and range of motion after coronary artery bypass grafting and concluded that the Pilates method is a safe, viable, and playful option for the patient profile after CABG but they did not evaluate kinesiophobia of patients

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable patient Who underwent elective CABG.
* Patients diagnosed with Kinesiophobia via Tampa scale for Kinesiophobia Heart (TSK-SV Heart)

Exclusion Criteria:

* Neuromuscular conditions which lead to kinesiophobia
* Diseases that seriously affected the functional capacity or mobility such as liver cirrhosis, chronic renal failure and disabled patients.
* Prolong intubation
* Vital instability
* Patients needing maximum assistance
* Decline consent

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | 2 weeks, 4 weeks
  Changes from baseline to 2 weeks and 4 weeks after intervention, measured through the TSK-SV Heart specifically focuses on assessing Kinesiophobia in the context of cardiac conditions or symptoms. It include questions related to fear of engaging in physical activity due to concerns about cardiac events (such as heart palpitations, chest pain, or shortness of breath) during exercise or daily activities. The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible Kinesiophobia, and the higher scores indicate an increasing degree of Kinesiophobia.
Abnormal heart rhythms | 2 Weeks, 6 Weeks
  Post-operative period and discharge day observed through Electrocardiography (ECG) on cardiac monitor.

SECONDARY OUTCOMES:
Functional mobility | 2 weeks, 4 weeks
  Changes from baseline to 2 weeks and 4 weeks after intervention, measured through the 10 meter walk test. It is a performance measure test used to assess walking speed in meters per second over a short distance . It can be employed to determine functional mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Lady Reading Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No